CLINICAL TRIAL: NCT04719325
Title: Comparative Study of Herbert Screw vs Lag Screw Fixation in Anterior Mandibular Fracture Treatment (a Clinical and Radiographic Study)
Brief Title: Herbert Screw vs Lag Screw Fixation in Anterior Mandibular Fracture Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hams Hamed Abdelrahman (Other)
Responsible Party: Sponsor-Investigator, Hams Hamed Abdelrahman, Assistant lecturer of DPH and Clinical statistician, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: herbert screw
Record Dates: First submitted 2021-01-17; First posted 2021-01-22 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Mandibular Fractures
MeSH Terms: conditions — Mandibular Fractures

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Herbert screw (Experimental)
  Interventions: Other: Herbert screw
- Lag screw (Active Comparator)
  Interventions: Other: Lag screw

INTERVENTIONS:
Other: Herbert screw — Fracture line exposed through intra-oral approach. bone reduction into proper anatomical occlusion and application of Herbert screw
  Arms: Herbert screw
Other: Lag screw — Fracture line exposed through intra-oral approach. bone reduction into proper anatomical occlusion. Application of either lag screw according to Champy's osteosynthesis lines.
  Arms: Lag screw

SUMMARY:
14 patients having recent anterior mandibular fracture divided into two groups. Group A has 6 patients and treated using Herbert bone screw, and group B has 6 patients and treated using lag screw.

Clinical follow-up was conducted after 24-hours, one, four, six, and twelve weeks. In addition, a radiographic investigation was performed after twelve weeks to estimate the mean bone density across the fracture line.

ELIGIBILITY:
Inclusion criteria

* Patients suffering from recent, uninfected anterior mandibular fracture.
* Adult patients from 20-60 years old with no gender predilection agreed to present for follow-up visits for a minimum postoperative period of 3 months.
* Fracture that demands open reduction and internal fixation.

Exclusion criteria

* Medically compromised patients contradicting operations.
* Existence of infection at the fracture line.
* Pathological fracture.
* An old fracture.
* Completely edentulous patient

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2019-10-18 (Actual); Primary Completion 2020-04-15 (Actual); Study Completion 2020-06-15 (Actual)

PRIMARY OUTCOMES:
Change in bone density | baseline and 3 months
  By using digital orthopantomogram bone density was evaluated
change in pain scores | 24 hours, 1 week , 4 Weeks and 6 weeks
  assessed through a 10-point Visual Analogue Scale (VAS). (0-1= None, 2-4= Mild, 5-7= Moderate, 8-10= Severe)
presence of Intra-fragmentary mobility | 24 hours
  assessed by bi-manual palpation across the fracture site

CONTACTS AND LOCATIONS:
Locations (1):
- Outpatient Clinic of Oral and Maxillofacial Surgery Department, Faculty of Dentistry, Alexandria University, Egypt, Alexandria, Azarita, Egypt